CLINICAL TRIAL: NCT00016926
Title: A Limited Access Phase II Trial Of Capecitabine In Advanced, Persistent Or Recurrent Squamous Cell Carcinoma Of The Cervix
Brief Title: Capecitabine in Treating Patients With Advanced, Persistent, or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068633; GOG-0076CC
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2004-05

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating patients who have advanced, persistent, or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of capecitabine in patients with advanced, persistent, or recurrent squamous cell carcinoma of the cervix.
* Determine the toxicity profile of this drug in this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 28-62 patients will be accrued for this study within 9-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced, persistent, or recurrent squamous cell carcinoma of the cervix

  * Documented disease progression after local therapy and considered incurable
* At least 1 target lesion measurable in at least 1 dimension

  * At least 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR at least 10 mm by spiral CT scan
  * Target lesion cannot be in a previously irradiated field

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine clearance at least 50 mL/min

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No neuropathy (sensory and motor) greater than grade I

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy or immunotherapy for the malignant tumor
* No concurrent prophylactic filgrastim (G-CSF)

Chemotherapy:

* At least 3 weeks since prior chemotherapy for the malignant tumor and recovered
* No prior cytotoxic therapy (except when used as a radiosensitizer)
* No prior chemotherapy for other malignancy

Endocrine therapy:

* At least 1 week since prior hormonal therapy for the malignant tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for the malignant tumor and recovered
* No prior radiotherapy for other malignancy

Surgery:

* Recovered from prior surgery

Other:

* At least 3 weeks since any other prior therapy for the malignant tumor
* No prior anticancer therapy that contraindicates study therapy
* No concurrent amifostine or other protective reagents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — University of Southern California
Locations (10):
- United States (9):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Garcia AA, Blessing JA, Darcy KM, Lenz HJ, Zhang W, Hannigan E, Moore DH. Phase II clinical trial of capecitabine in the treatment of advanced, persistent or recurrent squamous cell carcinoma of the cervix with translational research: a gynecologic oncology group study. Gynecol Oncol. 2007 Mar;104(3):572-9. doi: 10.1016/j.ygyno.2006.09.002. Epub 2006 Oct 17. PMID 17049588